CLINICAL TRIAL: NCT00742378
Title: Discriminating Ability of the Cirrus HD OCT for Glaucoma
Brief Title: Discriminating Ability of the Cirrus High Definition (HD) Optical Coherence Tomography (OCT) for Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Gong Je Seong, Yonsei University College of Medicine
Other Study IDs: 3-2008-0076-Reproducibility
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Retinal nerve fiber layer; Cirrus OCT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- C: Normal controls
- G: Glaucoma

SUMMARY:
The Cirrus HD OCT, a new spectral domain optical coherence tomography, has better resolution than the previous OCT. Reproducibility and discriminating ability of the Cirrus HD OCT for glaucoma detection will be studied.

DETAILED DESCRIPTION:
The Cirrus HD OCT is a newly developed imaging device of the spectral domain optical coherence tomography. Even though its resolution and speed are much better than the previous OCT, its reproducibility and diagnostic power for detecting the glaucomatous defect of retinal nerve fiber layer (RNFL) have not known yet. In the present study, we will review the data of RNFL thickness measurement using the Cirrus HD OCT. After assessing the inter-test variability, the discriminating ability of the Cirrus HD OCT for glaucoma diagnosis will be determined by the ROC curves.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative patients
* Repeated OCT data

Exclusion Criteria:

* Intraocular surgeries history
* DM
* High refractive error ( < -4.00 diopters, or > + 4.00 diopters)
* Media opacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients and normal controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-10 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness | when the OCT images are taking

SECONDARY OUTCOMES:
Red-free fundus photo | when the OCT images are taking
Visual field | when the OCT images are taking
Intraocular pressure | when the OCT images are taking

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Gong Je Seong, Seoul, South Korea